CLINICAL TRIAL: NCT03256760
Title: Experimental Model of Depression in Aging: Insomnia, Inflammation, and Affect Mechanisms
Brief Title: Sleep and Healthy Aging Research for Depression (SHARE-D) Study
Acronym: SHARE-D
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Irwin, MD (Other)
Responsible Party: Sponsor-Investigator, Michael Irwin, MD, Principal Investigator, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 16-000583
Record Dates: First submitted 2017-08-11; First posted 2017-08-22 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Depression in Old Age
Keywords: Insomnia, depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Endotoxins

STUDY DESIGN:
Intervention Model Description: Endotoxin vs. Placebo
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinded infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Endotoxin (Experimental): Endotoxin 0.8 ng/kg body weight
  Interventions: Biological: Endotoxin
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Endotoxin — Endotoxin
  Arms: Endotoxin
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Late-life depression is a significant public health concern, and effective interventions for prevention and treatment are needed. Insomnia and inflammation are modifiable targets for depression prevention, and this study is significant in using an experimental approach (i.e., inflammatory challenge) to probe acute inflammatory- and depression responses as a function of insomnia, which will inform identification of molecular targets for pharmacologic interventions, and improvement of insomnia treatments to prevent depression in older adults.

Project

DETAILED DESCRIPTION:
This study (SHARE-D) will use an inflammatory challenge (i.e., endotoxin) to probe acute inflammatory- and depression responses (primary outcome) in older adults as a function of insomnia. Older adults with insomnia show chronic inflammation; sleep disturbance also activates inflammatory signaling; chronic inflammation primes acute inflammatory responses; chronic inflammation, as well as acute inflammatory reactivity, predict depression over the following year; and finally, endotoxin induces acute inflammation along with depressive symptoms, with preliminary evidence that "two-hits" (i.e., sleep disturbance and inflammatory challenge) are associated with exaggerated increases in depression, especially in women. In this placebo-controlled, randomized, double-blind study of low dose endotoxin in older adults (60-80 y; stratified by sex) with insomnia (n=60) vs. comparisons without insomnia (n=100), the investigators hypothesize that older adults with insomnia will show heightened inflammatory- and affective responding to inflammatory challenge as compared to those without insomnia. The investigation aims to: 1) examine differences in depressive symptoms and measures of negative affect responding as a function of insomnia and inflammatory challenge; 2) examine differences in measures of positive affect responding as a function of insomnia and inflammatory challenge; and 3) examine differences in experimentally-induced inflammation in relation to depressive symptoms and measures of negative- and positive affect responding as a function of insomnia.

ELIGIBILITY:
* Inclusion Criteria:

  * Participants will be required to be in good general health (as evaluated during the phone and in-person baseline session)
  * Participants will be aged 60 to 80 years.
  * Half the participants (N=80) will be those with insomnia disorder as diagnosed by the Structured Clinical Interview for Diagnosis, Diagnostic Statistical Manual 5 and the Duke Structured Interview for Sleep Disorders, .
  * The other half will be those without insomnia identified as not having insomnia by any of these assessments.
* Exclusion Criteria: Following a structured telephone interview, prospective participants with the following conditions will not advance to the in-person baseline session:

  * Presence of chronic mental or physical illness (except for insomnia)
  * History of allergies, autoimmune, liver, or other severe chronic diseases,
  * Current and regular use of prescription medications such as steroids, non-steroid anti-inflammatory drugs, aspirin, immune modifying drugs, opioid analgesics, statins, antihypertensive drugs, anti-arrhythmic drugs, and antidepressant medications (none in the last 6 months); and nightshift work or time zone shifts (> 3hrs) within the previous 6 weeks, or previous history of fainting during blood draws.
  * Presence of co-morbid medical conditions not limited to but including cardiovascular (e.g., history of acute coronary event, stroke) and neurological diseases (e.g., Parkinson's disease), as well as pain disorders;
  * Presence of comorbid inflammatory disorders such as rheumatoid arthritis or other autoimmune disorders;
  * Presence of an uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or to put the study participant at undue risk;
  * Presence of chronic infection, which may elevate proinflammatory cytokines;
  * Presence of an acute infectious illness in the two weeks prior to an experimental session.
  * Current Axis I psychiatric disorders as determined by the Research Version of the Structured Clinical Interview including a current major depressive disorder and substance dependence (a prior history of depression is not an exclusion criterion, which will be considered for a pre-planned sensitivity analysis and will be used as a pre-classification variable in the generation of the two groups, and in the randomization schedule);
  * Lifetime history of suicide attempt or inpatient psychiatric admission. Sleep Disorders:
  * Current history of sleep apnea or nocturnal myoclonus;
  * Phase-shift disorder, which will be identified by the Structured Clinical Interview and the Duke Structured Interview for Sleep Disorders ; Medication and Substance Use:
  * Current and/or past regular use of hormone-containing medications including steroids;
  * Current and/or past regular use of non-steroid anti-inflammatory drugs;
  * Current and/or past regular use of immune modifying drugs that target specific immune responses such as cytokine antagonists;
  * Current and/or past regular use of analgesics such as opioids;
  * Current and/or past regular use of cardiovascular medications, including antihypertensive, antiarrhythmic, antianginal, and anticoagulant drugs;
  * Use of antidepressant medications or other psychotropic medications; (16) current smoking or excessive caffeine use (>600 mg/day) because of the known effects on proinflammatory cytokine levels;
  * Evidence of recreational drug use from urine test. Health Factors:
  * Body mass index > 35 because of the effects of obesity on proinflammatory cytokine activity and also on risk for sleep disordered breathing;
  * Any clinically significant abnormality on screening laboratory tests
  * Clinically significant abnormalities in electrocardiogram

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Depressed Mood Subscale of the Profile of Mood States (POMS) | 12 hours
  The Depressed Mood Subscale of the POMS is a self-and observer rated assessment of depressed mood in which severity of depressed mood is rated using a visual analog scale from 1 to 5 (5 being most severe). Each timepoint is scored and analyses examine the temporal profile of change with assessment every hour
Depressed mood and depressive symptoms as measured by the Montgomery Asberg Depression Rating Scale (MADRS) | 8 hours
  Depressed mood and depressive symptom severity by self-reported assessment using the Montgomery Asberg Depression Rating scale with a range from 0 to 54 with a higher score indicating more severe depressive symptoms. Each timepoint is scored and analyses examine the temporal profile of change with assessment every 2 hours

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | 8 hours
  The Hamilton Depression Rating Scale is on the most widely used scales in depression, which is adapted to evaluate acute changes in depressive symptoms. A trained interviewer, blind to the experimental condition, make ratings of items of depressed mood, feelings of guilt, loss of interest, retardation/agitation, anxiety, and somatic symptoms using items from the Hamilton Depression Rating Scale. The 17-item version will be used.
Emotion Facial Recognition Task | about 2 hours
  This is a computer-based test that includes color photographs of facial expression of evoked-or felt-emotions: happy, sad, angry, fearful, disgusted, and nonemotional or neutral. Participants rate the emotional valence using a scale of 0-8 of each expression.
Emotion Intensity Task | about 2 hours
  This is a computer-based test used along with emotion facial recognition to test subjective ratings of perceived intensity in response to facially-expressed emotions
Probabilistic Reward Task | about 2 hours
  This is a probabilistic reward task that is administered using computerized reward-learning task rooted in signal detection theory that yields an objective measurement of participant's ability to modulate behavior as a function of rewards. The variable that will be scored is termed response bias (RB), which reflects participants' preference for the stimulus paired with more frequent rewards.
Effort Expenditure for Reward Task | about 2 hours
  Similar to the Reward Learning Task, this is a computer based reward task to evaluate reward processing in the context of monetary reward.
Social Reward Task | about 2 hours
  This will evaluate another component of reward by subjective reports and task sensitivity to general social rewards
Snaith-Hamilton Pleasure Scale | 8 hours
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a self-administered questionnaire with 14 items assessing four domains of pleasure response/hedonic experience: interest/pastimes, social interaction, sensory experience, and food/drink, with each item scored from 1 to 4.
Temporal Experience of Pleasure Scale | 8 hours
  This self-report scale rates interest in 10 different activities, how much a person is interested in doing that activity right now

OTHER OUTCOMES:
Feelings of Social Disconnection | 12 hours
  Using the Feelings of Social Disconnection Scale, participant rated the extent to which they were feeling the ''following feelings right now" on a 5-point Likert scale (1-not at all, to 5- very much so): (1) ''I feel like being around other people," (2) ''I feel like being alone," (3) ''I feel overly sensitive around others (e.g., my feelings are easily hurt)," (4) ''I feel connected to others," and (5) ''I feel disconnected from others." Items 1 and 4 were reverse-coded, and scores were averaged at each time point to create a measure of self-reported social disconnection. Each timepoint is scored and analyses examine the temporal profile of change with assessment every hour
Physical symptoms | 12 hours
  Physical "sickness" symptoms which have been related to the administration of endotoxin are assessed during the experimental protocol; these sickness symptoms include self-reported rating of severity of muscle pain, shivering, nausea, breathing, difficulties, and fatigue
Psychiatric symptoms | 6 hours
  The Brief Symptom Inventory will be used assesses a wide variety of psychiatric symptoms
Systemic marker of inflammation as indexed by interleukin-6 | 12 hours
  Systemic inflammation as measured by circulating levels of interleukin-6 in plasma in pg/ml. Each timepoint is assayed and analyses examine the temporal profile of change with assessment every hour
Genomic marker of inflammation | about 2 hours
  Transcriptional profile of inflammation as measured by Conserved Translational Response to Adversity in circulating peripheral blood mononuclear cells
UCLA Loneliness Scale | 6 hours
  UCLA Loneliness scale is a 10-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as either O ("I often feel this way"), S ("I sometimes feel this way"), R ("I rarely feel this way"), N ("I never feel this way").
Social Status | 6 hours
  MacArthur Scale of Subjective Social Status (i.e., Social Ladder) will be used to evaluate perceived social status
Perceived Social Support | 6 hours
  Social Support Questionnaire Scale will be used to evaluated perceived social support
Social Attachment | 6 hours
  The Attachment Style Questions will be used to evaluate feelings of social attachment. This scale is reported 18 items that rates how you feel generally experience in relationships, not just in what is happening in a current relationship.
Sensitivity to Social Rejection | 6 hours
  Sensitivity to social rejection is examined by Fear of Negative Evaluation Scale and Mehrabian Rejection Sensitivity Scale
Cyberball Social Exclusion Task | 2 hours
  The Cyberball Social Exclusion Task is a virtual ball-toss game in which a participant plays with two other players (virtual) on a computer. Abruptly, the others exclude the participant, only throwing to one another. After completion of the task, the degree of perceived ostracism was was evaluated by a 20-item ostracism distress or social exclusion scale.
Cognitive Processing | 5.5 hours
  Increasing evidence indicates that inflammatory challenge acutely alters measures of cognitive performance, including spatial learning and memory. We use a virtual Morris Water Maze task (REF: https://pubmed.ncbi.nlm.nih.gov/19121374/) to assess computerized spatial learning and memory, followed by a Room Reconstruction Task (REF: https://pubmed.ncbi.nlm.nih.gov/10779831/) to assess the ability of cognitive mapping under real-life conditions.
Mechanical Temporal Summation | 5.5. hours
  Temporal summation reflects the endogenous capacity to enhance pain and will be assessed by calculating the windup ratio as a primary outcome for SHARE-Pain (or SHARE-P). Higher values are indicative of greater pain facilitation. Multiple pinprick probes were used (#3, #5, #6, and #7). The windup ratio will be calculated and z-scored within each probe. The z-scored windup ratios will then be averaged across probes to create an aggregate temporal summation index. Change scores will also be used to calculate temporal summation by subtracting the peak pain rating during 10 successive pinpricks from the pain rating during a single pinprick. The change scores will also be z-scored and averaged across probes. The windup ratio will be a primary outcome, whereas the change score metric will be a secondary outcome for SHARE-P.
Conditioned Pain Modulation | 5.5 hours
  Conditioned pain modulation assesses the degree to which one noxious stimulus reduces pain produced by a second noxious stimulus and is a measure of endogenous capacity for pain inhibition. It is calculated by taking the percent change in pressure pain threshold during the cold pressor task compared to the pressure pain threshold assessed just prior to cold water submersion. Larger values indicate better pain inhibitory capacity. This variable is a primary outcome for the SHARE-P. Raw difference scores will also be reported as a secondary outcome.
Affective Pain Modulation | 5.5
  Affective pain modulation refers to the ability of negative emotions to enhance pain while positive emotions reduce pain. Participants will be asked to rate their pain on a 0 (no sensation) to 100 (intolerable) scale to two thermal stimuli (46°C and 48°C) presented in a randomized order throughout each condition.Self-reported pain will be compared across the three conditions (negative, positive, neutral). Affective pain modulation is a primary outcome for SHARE-
Pressure Pain Threshold-Trapezius muscle | 5.5 hours
  Pressure pain threshold is the pressure that first elicits pain, such that lower values indicate greater pain sensitivity. Pressure pain threshold was assessed at three sites: trapezius, masseter, and middle insertion of the quadriceps. Four trials were completed at each site (two on the left side two on the right side). All threholds will be z-scored within each site and averaged across sites to create an index score. Pressure pain threshold is a secondary outcome for SHARE-P.
Heat Pain Threshold | 5.5 hours
  The first thermal stimulus that participants self-report as painful (averaged across two trials). Lower values indicate enhanced pain sensitivity. This is a secondary outcome variable for the SHARE-P sub-study.
Heat Pain Tolerance | 5.5 hours
  The thermal stimulus at which the participant identifies the pain as intolerable (averaged across two trials). Lower values represent greater pain sensitivity. This is a secondary outcome variable for the SHARE-P sub-study.
Cold Pain Tolerance | 5.5
  Cold pain tolerance is measured as the time it takes for the participant to withdraw their hand from cold water bath (2°C), such that shorter durations reflect greater pain sensitivity. (Secondary outcome for SHARE-P).
Pain Pain Threshold. Masseter muscle and middle of quadriceps | 5.5 hours
  * Pressure pain threshold is the first mechanical stimulus that a participant self-reports as painful, such that lower values indicate greater pain sensitivity. Pressure pain threshold is the average of two readings and will be reported separately for the masseter muscle and middle of the quadriceps. These are tertiary outcomes for SHARE-P.
Pain Intensity | 12 months
  Pain intensity ratings will be assessed daily using a Visual Analogue Scale and averaged across the two week period to determine the Pain Intensity Index. These ratings will be made at baseline, 3mo, 6mo, 9mo, and 12mo and are considered a primary outcome for the longitudinal component of SHARE-P.
Depressive symptoms | 12 months
  Depressive symptoms will be assessed at baseline, 3mo, 6mo, 9mo, and 12mo using the Patient Health Questionnaire - 9 item (PHQ-9). This is a primary outcome for the longitudinal component of SHARE-P.
Graded Chronic Pain Scale | 12 months
  Pain intensity and pain-related disability are assessed at baseline, 3mo, 6mo, 9mo, and 12mo using the Graded Chronic Pain Scale (3-month version). This is a secondary outcome for the SHARE-P study.
Affective Disturbance | 12 months
  o Affective disturbance is assessed daily during a 2-week period by having participants rate the extent to which they feel three positive (happy, calm, agreeable) and three negative emotions (sad, anxious, annoyed) on a 0 (not at all) to 100 (extremely) scale. Daily positive affect and negative affect are calculated by averaging across the three positive and negative emotion words, respectively. Participants complete these measures at baseline, 3mo, 6mo, 9mo and 12mo. This is a secondary outcome for SHARE-P.
Sleep Continuity | 12 months
  Electronic sleep diaries will be administered daily for two weeks at baseline, 3mo, 6mo, 9mo, and 12mo. Sleep diaries will be used to assess sleep continuity, including (1) latency to initial sleep onset, (2) frequency of nightly awakenings, (3) wake after sleep onset, (4) total sleep time, and (5) sleep efficiency (total sleep time/time in bed). These are considered secondary outcomes for SHARE-P.
Total Sleep Time | 12 months
  Participants will receive an ActiGraph (wrist triaxial accelerometer) to wear for a 2-week period at baseline, 3mo, 6mo, 9mo, and 12mo to measure total sleep time (secondary outcome for SHARE-P).

CONTACTS AND LOCATIONS:
Locations (1):
- Cousins Center for Psychoneuroimmunology, UCLA Neuropsychiatric Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after study completion
Access Criteria: Contact PI to obtain permission for data release

REFERENCES:
- [Derived] Boyle CC, Cho JH, Eisenberger NI, Olmstead R, Sadeghi N, Castillo D, Irwin MR. Inflammation-induced depressed mood and reward responsivity as a function of age in female adults: a randomized controlled trial of endotoxin. Transl Psychiatry. 2025 Nov 26;16(1):6. doi: 10.1038/s41398-025-03752-2. PMID 41298372
- [Derived] Irwin MR, Boyle CC, Cho JH, Piber D, Sadeghi N, Castillo D, Smith MT, Eisenberger NI, Olmstead R. Inflammatory Exposure and Depression in Older Adults With Insomnia: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Sep 1;82(9):859-867. doi: 10.1001/jamapsychiatry.2025.1327. PMID 40668551
- [Derived] DuPont CM, Olmstead R, Reid MJ, Hamilton KR, Campbell CM, Finan PH, Sadeghi N, Castillo D, Irwin MR, Smith MT. A randomized, placebo-controlled, double-blinded mechanistic clinical trial using endotoxin to evaluate the relationship between insomnia, inflammation, and affective disturbance on pain in older adults: A protocol for the sleep and Healthy Aging Research for pain (SHARE-P) study. Brain Behav Immun Health. 2023 May 19;30:100642. doi: 10.1016/j.bbih.2023.100642. eCollection 2023 Jul. PMID 37256193